CLINICAL TRIAL: NCT07196553
Title: Role of Ultrasound in Ascites: Detection, Characterization, and Evaluation of the Underlying Cause.
Brief Title: Ultrasound and Ascites
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Sayed Abdelaziz, Dr, Assiut University
Other Study IDs: Role of ultrasound in ascites
Record Dates: First submitted 2025-09-13; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ultrasound in Ascites
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — ultrasound examination

SUMMARY:
The aim of this study is to evaluate the role of ultrasound in the detection, characterization, and determination of the underlying cause of ascites in patients attending Assiut University Hospital

DETAILED DESCRIPTION:
Normally, the peritoneal cavity contains 25-50 mL of ascitic fluid, which allows for the movement of bowel loops past one other and helps hydrate serosal surfaces. Ascites is defined as the pathological accumulation of excess fluid in the peritoneal cavity.

More than one cause may be responsible for the development of ascites (multifactorial), liver cirrhosis remains the leading cause (≈85% of cases), followed by many causes such as malignant neoplasia, tuberculous infection, cardiac insufficiency, renal diseases ,trauma and other infectious, inflammatory and hemorrhagic causes ,multiple etiologies may coexist.

once ascites develops, it carries a risk of further serious complications such as acute spontaneous bacterial peritonitis (SBP) (Occurs in 10-30% of hospitalized cirrhotic patients with ascites and associated with high morbidity and mortality rate), hepatorenal syndrome, hepatic hydrothorax, respiratory compromise and other compliactions including gastrointestinal, circulatory , metabolic complications….etc Medical history, physical examination, abdominal ultrasound, blood tests, and a diagnostic paracentesis for ascitic fluid analysis should all be part of the initial assessment of ascites. Ascites can be detected on physical examination using traditional shifting dullness to percussion when there is approximately 500 ml of fluid. However, in an increasingly obese population, there is limited reliability on clinical examination findings alone.

Trans-abdominal US (TAUS) can easily demonstrate large volumes of fluid and, with a meticulous technique, much smaller volumes can also be detected making an excellent first-line imaging tool, safe, inexpensive, and widely available, It's also superior to CT in qualitative assessment-distinguishing between simple (anechoic) and complex (particulate or septated) ascites.Portable ultrasound devices further enable reliable, bedside diagnosis.

Ultrasound is also used in ultrasound-guided aspiration and paracentesis which is essential for safely obtaining ascitic fluid for determining the underlying etiology (via Serum-Ascites Albumin Gradient (SAAG), cytology, biochemical analysis) and detecting complications such as spontaneous bacterial peritonitis,The presence of septations or debris in ascites fluid can be suggestive of infected ascites.

The most important diagnostic study of any patient being evaluated for SBP or being admitted to the hospital with ascites and cirrhosis is a paracentesis. In a US national inpatient study of over 31,000 patients admitted with cirrhosis and ascites where about one-half underwent a paracentesis, the mortality rate for patients who underwent a paracentesis was significantly lower than for those who did not have one (6.3% vs 8.9%). hemorrhagic ascites, or malignant recurrence.

Real-time ultrasound improves diagnostic accuracy and reduces complication rates compared with landmark-based aspiration..Using ultrasound guidance for paracentesis significantly reduces complication rates, such as bleeding and infection.complication rates drop from ~4.7% (landmark-based) to ~1.4% with ultrasound.

therapeutic paracentesis is established as the first-line treatment for patients with large or refractory ascites providing rapid symptom relief and improving quality of life. It is safe when done under ultrasound guidance with albumin replacement for large-volume drainage.

' We chose to carry out this study to evaluate the specificity, sensitivity, accuracy, and positive and negative predictive value of role of ultrasound in detection of ascites and evaluation of the underlying cause.

ELIGIBILITY:
Inclusion Criteria:

* Patient from different age groups and both sexex will be included in our study.
* Patients with clinically suspected ascites referred for abdominal ultrasound.
* Patients who will provide informed consent for participation.

Exclusion Criteria:

* Patients with a history of recent abdominal surgery (<1 month).
* Patients with inadequate ultrasound visualization due to severe obesity or extensive bowel gas.
* Patients who will decline to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: -Patients attending Assiut University Hospital from different age groups and both sexex with clinically suspected ascites referred for abdominal ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Role of ultrasound in ascites | Baseline
  To evaluate the accuracy of ultrasound in ascites detection and characterization.

OTHER OUTCOMES:
role of ultrasound in ascites | Baseline
  to evaluate the role of ultrasound in the detection, characterization, and determination of the underlying cause of ascites in patients attending Assiut University Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sami Abdel-Aziz Khalil, proffesor, Study Director — Assiut University